CLINICAL TRIAL: NCT06450067
Title: To Observe and Evaluate the Efficacy and Safety of Inaticabtagene Autoleucel Injection in the Treatment of Relapsed or Refractory B-cell Acute Lymphoblastic Leukemia in Adults in the Real World
Brief Title: Inaticabtagene Autoleucel Injection Treatment for Adult Relapsed or Refractory Acute Lymphocytic Leukemia
Status: Recruiting | Type: Observational
Sponsor: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: HY001402
Record Dates: First submitted 2024-06-03; First posted 2024-06-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnosed relapsed or refractory B-cell acute lymphoblastic leukemia: Diagnosed relapsed or refractory B-cell acute lymphoblastic leukemia

SUMMARY:
This clinical trial is a non-interventional, observational, multicenter, post-marketing real-world study to evaluate the efficacy and safety of Inaticabtagene Autoleucel Injection in Chinese adult patients with relapsed or refractory B-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
The study is a non-interventional, observational, multicenter, post-marketing real-world study, and its objective is to evaluate the efficacy and safety of Inaticabtagene Autoleucel Injection in the treatment of Relapsed or Refractory acute lymphoblastic leukemia. The study consists of screening period including leukapheresis, treatment period, and follow-up period (2 years at most).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Diagnosed with relapsed or refractory B-cell acute lymphoblastic leukemia;
3. Patients deemed eligible for receiving commercial Inaticabtagene Autoleucel injection treatment as determined by the investigator;
4. Patients voluntarily participate in this study and sign an informed consent form. For patients lacking full legal capacity, informed consent must be obtained from their legal guardian

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed with adult relapsed or refractory B-cell acute lymphoblastic leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2029-06-05 (Estimated)

PRIMARY OUTCOMES:
overall survival | 2 years
  OS is defined as the time from the start date of Inaticabtagene Autoleucel Injection infusion to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China; Aibin Liang, Dr., Principal Investigator — Tongji Hospital
Locations (10):
- China (10):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Henan Cancer Hospital Affiliated Cancer Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Qilu Hospital of Shandong university, Jinan, Shandong
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - West China School of Medicine/West China Hospital of Sichuan University, Chengdu, Sichuan
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No